CLINICAL TRIAL: NCT03187587
Title: An Open-Label, Comparative Trial to Evaluate the Effect of imILT in Patients With Advanced Disease or Stage IV Pancreatic Carcinoma
Brief Title: Percutaneous Immunostimulating Interstitial Laser Thermotherapy in Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped in agreement with investigator due to slow recruitment.
Sponsor: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2015-006
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms Pancreatic
Keywords: Hyperthermia, Induced; Laser Coagulation; Laser Therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- imILT treatment (Experimental): Immunostimulating Interstitial Laser Thermotherapy (imILT)
  Interventions: Device: imILT
- Standard chemotherapy treatment (Active Comparator): This study arm recieves chemotherapy treatment as standard care at the clinical study site.
  Interventions: Drug: Standard chemotherapy treatment

INTERVENTIONS:
Device: imILT — The imILT treatment arm recieves imILT treatment and no simultaneous chemotherapy.
  Other Names: TRANBERG Thermal Therapy System
  Arms: imILT treatment
Drug: Standard chemotherapy treatment — The standard chemotherapy treamtment arm recieves only chemotherapy.
  Arms: Standard chemotherapy treatment

SUMMARY:
Thermotherapy is a technology aiming at destroying tissue, for example tumor tissue. Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response. In laboratory animals the imILT method has also been shown to induce a so called abscopal effect. This means that when one tumor is treated with imILT other, untreated, tumors also decrease in size.

The purpose of this trial is to evaluate efficiency when it comes to local tumor destruction of the imILT treatment method performed pecutaneously in patients diagnosed with pancreatic cancer. The purpose is also to investigate the functionality and safety of the method.

This trial is an open-label, double-arm study. Twenty patients diagnosed with pancreatic cancer will be treated in this trial, ten recieving imILT treatment and ten recieving standard chemotherapy. The study is estimated to be carried out during a time period of 21 months.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of non-resectable pancreatic adenocarcinoma by form of either locally advanced disease (stage II-III) or of stage IV disease with hepatic metastasis (staging according to UICC 2009)
* Locally advanced disease shall have a lesion diameter less than 4cm
* If stage IV disease, the patient shall have only liver metastasis, with less than 5 in number, each one less than 4 cm in diameter
* The patient is a candidate for standard chemotherapy (as described at point 5.1)
* Age between 18 and 80 years, males and females
* Anticipated compliance with treatment and follow-up
* Have given informed verbal and written consent to participation in the trial
* Have stable and adequate haematologic, renal and hepatic functions:

  1. Hemoglobin ≥9 g/dL
  2. Platelet count ≥75 x 109/L
  3. International normalized ratio (INR) ≤1.7
  4. WBC count ≥2 x 109/L
  5. Absolute neutrophil count (ANC) ≥1 x 109/L
  6. Albumin ≥2.8 g/dL, total bilirubin ≤3.0 mg/dL (51.3 μmol/L); ALT, AST ≤5 times upper limit of normal (ULN)
  7. Serum chemistries sodium, potassium, and calcium within normal limits (WNL)
  8. Serum creatinine <2.0 mg/dL or creatinine clearance >60 mL/min according to Cockroft-Gault formula
* At least a part of the tumour can be treated with imILT without damage to adjacentvital structures
* Have an ECOG performance status <2 (Karnofsky> 60%)

Exclusion Criteria:

* HIV 1 or 2 positive
* Active autoimmune disease which is judged to reduce an anti-tumour immune response
* Pregnancy or breast feeding
* Have known bleeding disorder that cannot be managed accordingly with the protocol rules, such severe acute or chronic liver failure, other genetic blood diseases not properly managed prior to treatment or other any disease treated with anticoagulant or anti-platelet medication that cannot be interrupted prior to treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment effect by radiology | 12 months
  Evaluation by Response Evaluation Criteria in Solid Tumours (RECIST)

SECONDARY OUTCOMES:
Safety assessed by the incidence the of adverse events | 12 months
  Evaluation of adverse events and laboratory analyses.
Usability (user evaluation of instrument) | 12 months
  Analysis of instrument and user questionnaires relating to the ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Belarmino Goncalves, MD, Principal Investigator — Portuguese Oncology Institute of Porto
Locations (1):
- Portuguese Oncology Institute of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No